CLINICAL TRIAL: NCT03932162
Title: Gene Expression Changes in Young and Geriatric Skin
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06694
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: UVB Phototherapy Burn; Insulin-like Growth Factor 1; Aging
MeSH Terms: interventions — Insulin-Like Growth Factor I

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Young Adult (Placebo Comparator): One small area of skin will undergo treatment with a small amount of UVB.
  Interventions: Other: No Insulin-Lie Growth Factor 1
- Geriatric Adult (Active Comparator): Four small areas will undergo injection of a small amount of IGF-1 drug and two will undergo injections with saline. Then the injected areas will be treated with a small amount of UVB.
  Interventions: Drug: Insulin-Like Growth Factor 1

INTERVENTIONS:
Drug: Insulin-Like Growth Factor 1 — Growth factor protein
  Arms: Geriatric Adult
Other: No Insulin-Lie Growth Factor 1 — No Insulin-Like Growth Factor 1 will be given.
  Arms: Young Adult

SUMMARY:
This study does not involve any particular diagnosis. The goal of this research study is to explore the effects of artificial sunlight (ultraviolet B radiation; UVB) on the skin of young adults versus geriatric adults. Sunlight exerts many effects on the body. There is evidence that in response to ultraviolet B radiation (UVB), which are the burning rays of sunlight, young adult skin responds differently than geriatric skin. In fact, researchers feel that this difference in how the skin reacts to UVB is why skin cancers are found in older skin. Researchers believe that a major difference between young adult and geriatric skin is that young skin has a lot of a protein called insulin-like growth factor-1 (IGF-1), whereas geriatric skin has very little. The current study will test how young adult versus geriatric skin responds to UVB, and if geriatric skin treated with an injection of small amount of IGF-1 drug will then act like young skin.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* White skin (Fitzpatrick types I and II)
* Age 21-30 or 65 and older
* Able to comprehend procedures/risks

Exclusion Criteria:

* Known photosensitivity
* Currently on photosensitizing medications
* Diabetes Mellitus
* History of abnormal scarring
* History of skin infections
* Known allergy to lidocaine local anesthetic
* Pregnancy or nursing
* Other serious health issues

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-09-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in expression genes involved in protecting skin cells from UVB damage in younger skin and geriatric skin injected with IGF-1 from baseline | 2 Days
  Expression genes involved in protecting skin cells from UVB damage, including p21, xeroderma pigmentosum (XPC), and polymerase eta, will be higher following UVB exposure in younger skin and geriatric skin injected with IGF-1 than in geriatric skin injected with saline as a control.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Travers, MD, PhD, Principal Investigator — Wright State University
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT03932162/ICF_000.pdf